CLINICAL TRIAL: NCT04599907
Title: An Evaluation of the Safety and Effectiveness of the N-SWEAT Patch for the Treatment of Primary Axillary Hyperhidrosis or Excessive Axillary Sweating
Brief Title: Evaluation of N-SWEAT Patch for Treatment of Primary Axillary Hyperhidrosis or Excessive Axillary Sweating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Candesant Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CB-CLP-001
Record Dates: First submitted 2020-10-06; First posted 2020-10-23 (Actual); Results first posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-08

CONDITIONS: Primary Axillary Hyperhidrosis
Keywords: Excessive Axillary Sweating; Primary Axillary Hyperhidrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Roll-In Cohort: N-SWEAT Patch (Experimental): Subjects will be treated with N-SWEAT Patch
  Interventions: Device: Roll-In Cohort: Single Application of N-SWEAT Patch
- Randomized Cohort: N-SWEAT Patch (Experimental): Subjects will be treated with N-SWEAT Patch
  Interventions: Device: Randomized Cohort: Single Application of N-SWEAT Patch
- Randomized Cohort: Sham Patch (Sham Comparator): Subjects will undergo identical procedure with an inactive sham device
  Interventions: Device: Randomized Cohort: Single Application of Sham Patch

INTERVENTIONS:
Device: Roll-In Cohort: Single Application of N-SWEAT Patch — Single Application of N-SWEAT Patch in both axillae for 10 subjects
  Arms: Roll-In Cohort: N-SWEAT Patch
Device: Randomized Cohort: Single Application of N-SWEAT Patch — Single Application of N-SWEAT Patch in both axillae for subjects randomized to the treatment group
  Arms: Randomized Cohort: N-SWEAT Patch
Device: Randomized Cohort: Single Application of Sham Patch — Single Application of Sham Patch in both axillae for subjects randomized to the control group
  Arms: Randomized Cohort: Sham Patch

SUMMARY:
The Sahara Study is a study to evaluate the safety and effectiveness of the N-SWEAT Patch for use in subjects with excessive axillary sweating, or primary focal axillary hyperhidrosis.

DETAILED DESCRIPTION:
The Sahara Study is intended to evaluate the safety and effectiveness of the N-SWEAT Patch for use in subjects with excessive axillary sweating, or primary focal axillary hyperhidrosis.

Safety of the N-SWEAT Patch will be confirmed by assessing the occurrence of local skin reactions, treatment-related adverse events (AEs) and Serious Adverse Events (SAEs).

Demonstration of effectiveness will be assessed by a significant improvement (reduction) in Hyperhidrosis Disease Severity Score (HDSS) in subjects treated with the N-SWEAT Patch. Secondary and additional endpoints based on complementary clinical instruments, including Quality of Life Measures (QOL) and Gravimetric Sweat Production GSP), have been included to further demonstrate performance.

ELIGIBILITY:
Key Inclusion Criteria:

1. Signed written informed consent
2. At least 22 years old at the time of consent.
3. Female or male, who experiences excessive sweating or has been diagnosed with primary axillary focal hyperhidrosis and is in otherwise good general health
4. GSP >50mg/5min in each axilla
5. Reports a score of HDSS score of 3 or 4

Key Exclusion Criteria:

1. Active skin disease, irritation, or abrasions at either axilla based
2. Subject's medical history is indicative of secondary or diffuse hyperhidrosis and/or subject has a diagnosis of secondary or diffuse hyperhidrosis
3. GSP exceeds 300 mg/5min in either axilla

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2021-07-06 (Actual); Study Completion 2021-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Walker, MD, Study Director — Candesant Biomedical - Medical Monitor
Locations (9):
- United States (9):
  - CA Dermatology & Clinical Research Inst, Encinitas, California
  - Center for Dermatology Clinical Research, Fremont, California
  - AE Derm, Rockville, Maryland
  - Skincare Physicians, Boston, Massachusetts
  - Grekin Skin Institute, Warren, Michigan
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Dermatology Consulting Services, Zoe Draelos, MD, High Point, North Carolina
  - Research Your Health, Dallas, Texas
  - Pariser Derm / Virginia Clinical Research, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Doolittle J, Walker P, Mills T, Thurston J. Hyperhidrosis: an update on prevalence and severity in the United States. Arch Dermatol Res. 2016 Dec;308(10):743-749. doi: 10.1007/s00403-016-1697-9. Epub 2016 Oct 15. PMID 27744497
- [Background] Glaser DA, Coleman WP 3rd, Fan LK, Kaminer MS, Kilmer SL, Nossa R, Smith SR, O'Shaughnessy KF. A randomized, blinded clinical evaluation of a novel microwave device for treating axillary hyperhidrosis: the dermatologic reduction in underarm perspiration study. Dermatol Surg. 2012 Feb;38(2):185-91. doi: 10.1111/j.1524-4725.2011.02250.x. Epub 2012 Jan 30. PMID 22289389
- [Background] Glaser DA, Hebert A, Pieretti L, Pariser D. Understanding Patient Experience With Hyperhidrosis: A National Survey of 1,985 Patients. J Drugs Dermatol. 2018 Apr 1;17(4):392-396. PMID 29601615
- [Background] Hamm H. Impact of hyperhidrosis on quality of life and its assessment. Dermatol Clin. 2014 Oct;32(4):467-76. doi: 10.1016/j.det.2014.06.004. Epub 2014 Jul 16. PMID 25152339
- [Background] Hornberger J, Grimes K, Naumann M, Glaser DA, Lowe NJ, Naver H, Ahn S, Stolman LP; Multi-Specialty Working Group on the Recognition, Diagnosis, and Treatment of Primary Focal Hyperhidrosis. Recognition, diagnosis, and treatment of primary focal hyperhidrosis. J Am Acad Dermatol. 2004 Aug;51(2):274-86. doi: 10.1016/j.jaad.2003.12.029. No abstract available. PMID 15280848
- [Background] Stander M, Wallis LA. The emergency management and treatment of severe burns. Emerg Med Int. 2011;2011:161375. doi: 10.1155/2011/161375. Epub 2011 Sep 4. PMID 22046536
- [Background] Strutton DR, Kowalski JW, Glaser DA, Stang PE. US prevalence of hyperhidrosis and impact on individuals with axillary hyperhidrosis: results from a national survey. J Am Acad Dermatol. 2004 Aug;51(2):241-8. doi: 10.1016/j.jaad.2003.12.040. PMID 15280843
- [Background] Wade R, Rice S, Llewellyn A, Moloney E, Jones-Diette J, Stoniute J, Wright K, Layton AM, Levell NJ, Stansby G, Craig D, Woolacott N. Interventions for hyperhidrosis in secondary care: a systematic review and value-of-information analysis. Health Technol Assess. 2017 Dec;21(80):1-280. doi: 10.3310/hta21800. PMID 29271741
- [Background] Wilke K, Martin A, Terstegen L, Biel SS. A short history of sweat gland biology. Int J Cosmet Sci. 2007 Jun;29(3):169-79. doi: 10.1111/j.1467-2494.2007.00387.x. PMID 18489347

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Roll-In Cohort: N-SWEAT Patch | Randomized Cohort: N-SWEAT Patch | Randomized Cohort: Sham Patch
Started | 10 (All outcomes were assessed by participant, both axilla were given the same treatment and the overall result for the patient was evaluated to determine safety and efficacy.) | 53 (All outcomes were assessed by participant, both axilla were given the same treatment and the overall result for the patient was evaluated to determine safety and efficacy.) | 57 (All outcomes were assessed by participant, both axilla were given the same treatment and the overall result for the patient was evaluated to determine safety and efficacy.)
Completed | 9 | 45 | 51
Not Completed | 1 | 8 | 6
Not completed — Withdrawal by Subject | 1 | 7 | 6
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Roll-In Cohort: N-SWEAT Patch | Randomized Cohort: N-SWEAT Patch | Randomized Cohort: Sham Patch | Total
Number analyzed (Participants) | 10 | 53 | 57 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 53 | 57 | 120
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.9 (15.3) | 32.6 (7.3) | 34.4 (8.4) | 34.3 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 30 | 36 | 73
  Male | 3 | 23 | 21 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 9 | 15
  Not Hispanic or Latino | 9 | 48 | 48 | 105
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 2 | 3
  Asian | 1 | 8 | 5 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 0 | 12 | 13 | 25
  White | 9 | 31 | 37 | 77
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 53 | 57 | 120
HDSS [Count of Participants; unit: Participants] — Hyperhidrosis Disease Severity Scale (HDSS) is a disease-specific diagnostic tool that provides a qualitative measure of the severity of the patient's condition based on how it affects daily activities. This study enrolled those with HDSS 3 or HDSS 4 only.
  1 - My sweating is never noticeable and never interferes with my daily activities 2- My sweating is tolerable but sometimes interferes with my daily activities 3- My sweating is barely tolerable and frequently interferes with my daily activities 4- My sweating is intolerable and and always interferes with my daily activities
  Participants
    HDSS 3 | 4 | 21 | 25 | 50
    HDSS 4 | 6 | 32 | 32 | 70

OUTCOME MEASURES:

1. Primary Outcome: Safety of the N-SWEAT Patch
Description: Number of patients with Adverse Events and/or Skin reactions following patch treatment
Time Frame: 4 weeks
Population: All subjects treated with the N-SWEAT Patch (roll-in and randomized) were combined into a single population for the safety analysis.
Measure: Count of Participants; unit: Participants
Groups:
- N-SWEAT Patch Treated: Subjects will be treated with N-SWEAT Patch
  Randomized Cohort: Single Application of N-SWEAT Patch: Single Application of N-SWEAT Patch in both axillae for subjects randomized to the treatment group
Arm/Group | N-SWEAT Patch Treated | Randomized Cohort: Sham Patch
Number analyzed (Participants) | 63 | 57
Participants | 14 | 4

2. Primary Outcome: Effectiveness of the N-SWEAT Patch to Change Subjects From an HDSS 3 or 4 at Baseline to HDSS 1 or 2 at 4 Weeks
Description: Achievement of Hyperhidrosis Disease Severity Scale (HDSS) score of 1 or 2 at 4 weeks.
  HDSS is a disease-specific diagnostic tool that provides a qualitative measure of the severity of the patient's condition based on how it affects daily activities. HDSS 3 or 4 are generally considered to have a clinically significant case and those with HDSS 1 or 2 are considered to have mild to no evidence of hyperhidrosis.
  SCALE: 1 - My sweating is never noticeable and never interferes with my daily activities 2- My sweating is tolerable but sometimes interferes with my daily activities 3- My sweating is barely tolerable and frequently interferes with my daily activities 4- My sweating is intolerable and and always interferes with my daily activities
Time Frame: 4 weeks
Population: This was conducted on the Efficacy Cohort which included only randomized/blinded subjects. Those treated in the roll-in cohort was not included in the efficacy analyses were aware of the treatment arm to which they were assigned. Additionally, subjects who were found to have been enrolled while taking a conflicting medication were excluded from the efficacy analysis in order to isolate the true device effect.
Measure: Count of Participants; unit: Participants
Groups:
- Randomized Cohort: N-SWEAT Patch Treated: Subjects will be treated with N-SWEAT Patch
  Randomized Cohort: Single Application of N-SWEAT Patch: Single Application of N-SWEAT Patch in both axillae for subjects randomized to the treatment group
Arm/Group | Randomized Cohort: N-SWEAT Patch Treated | Randomized Cohort: Sham Patch
Number analyzed (Participants) | 44 | 43
Participants | 28 | 19
Statistical Analysis 1: Comparison: Randomized Cohort: N-SWEAT Patch Treated vs Randomized Cohort: Sham Patch; Test type: Superiority; p < 0.05, Cochran-Mantel-Haenszel

3. Secondary Outcome: Mean Change in the Quality of Life. Assessed by Evaluating How Much Sweat Bothers or Impacts the Daily Life of Patients (a Higher Score Means More Bother and More Impact)
Description: Two Quality of Life (QoL) Assessments were conducted as part of this endpoint. The Level of Bother: Subjects were asked how much their sweat bothered them on a Scale of 1 (not at all bothered by sweating) to 5 (extremely bothered by sweating). The Impact of Sweat on Daily Activities: Subjects were asked how much their sweating impacts their daily activities on a scale of 1 (not at all impacted) to 5 (extremely impacted).
  The mean improvement of each of these was calculated by comparing the mean baseline level to the mean level at 4 weeks. The mean change in the level of improvement was analyzed for significance. A larger decrease in these levels, i.e. less bother and less impact, (indicated by a larger negative number) will show the most improvement in QoL.
Time Frame: 4 weeks
Population: The efficacy population was defined in efficacy primary outcome section. It included randomized subjects who were not taking any conflicting medications.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Randomized Cohort: N-SWEAT Patch Treated | Randomized Cohort: Sham Patch
Number analyzed (Participants) | 44 | 43
score on a scale
  Change in the Level of Bother due to Sweat | -1.52 [-1.88 to -1.16] | -0.61 [-0.98 to -0.25]
  Change in Level of Impact of Sweat on Daily Activities | -1.44 [-1.77 to -1.10] | -0.57 [-0.91 to -0.23]
Statistical Analysis 1: Comparison: Randomized Cohort: N-SWEAT Patch Treated vs Randomized Cohort: Sham Patch; This is the data for the "Level of Bother"statistical analysis; Test type: Superiority; p < 0.05, Mixed Models Analysis; Mean Difference (Final Values) = -0.91, 95% CI 2-sided [-1.42 to -0.040]
Statistical Analysis 2: Comparison: Randomized Cohort: N-SWEAT Patch Treated vs Randomized Cohort: Sham Patch; This is the data for the "Level of Impact on Daily Activities" Statistical Analysis; Test type: Superiority; p < 0.05, Mixed Models Analysis; Mean Difference (Final Values) = -0.87, 95% CI 2-sided [-1.35 to -0.40]

4. Secondary Outcome: Percentage of Patients With a Mean Change in Gravimetric Sweat Production (GSP) Indicating That Sweating After Treatment is Cut in Half From Pre-treatment Sweat
Description: Gravimetric Sweat Production (GSP) measures the amount of sweat that is produced in a 5-minute period. The percentage of treated subjects with at least a 50% reduction in mean GSP (mean of both axilla) from baseline to 4 weeks was analyzed for this endpoint.
Time Frame: 4 weeks
Population: This endpoint defined by the study protocol was for at least 50% of the treated subjects to achieve a reduction in GSP of 50% or more, thus, the sham population was not included in this analysis. Moreover, the GSP measurement (unlike the HDSS or the QoL measurements) required the subjects to report back to the clinic at 4-weeks. Only 43 of the 44 N-SWEAT treated subjects in the efficacy population reported for the 4-week visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Cohort: N-SWEAT Patch Treated
Number analyzed (Participants) | 43
Participants | 26

5. Secondary Outcome: Percentage of Patients With a 2-point Change in HDSS to Show That Sweat is Less Clinically Significant After Treatment
Description: Patients with a 2-point decrease in HDSS indicate improvement in sweating.
  HDSS is a disease-specific diagnostic tool that provides a qualitative measure of the severity of the patient's condition based on how it affects daily activities. HDSS 3 or 4 are generally considered to have a clinically significant case and those with HDSS 1 or 2 are considered to have mild to no evidence of hyperhidrosis.
  SCALE: 1 - My sweating is never noticeable and never interferes with my daily activities 2- My sweating is tolerable but sometimes interferes with my daily activities 3- My sweating is barely tolerable and frequently interferes with my daily activities 4- My sweating is intolerable and always interferes with my daily activities
Time Frame: 4-weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Cohort: N-SWEAT Patch Treated | Randomized Cohort: Sham Patch
Number analyzed (Participants) | 44 | 43
Participants | 19 | 7

ADVERSE EVENTS:
Time Frame: Adverse Events were collected for 12 weeks, the total duration of the study
Description: Definitions were consistent with clinicaltrials.gov.
Groups:
- N-SWEAT Patch: Subjects will be treated with N-SWEAT Patch
  Single Application of N-SWEAT Patch: Single Application of N-SWEAT Patch in both axillae for subjects randomized to the treatment group
- Sham Patch: Subjects will undergo identical procedure with an inactive sham device
  Randomized Cohort: Single Application of Sham Patch: Single Application of Sham Patch in both axillae for subjects randomized to the control group
Arm/Group | N-SWEAT Patch | Sham Patch
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/57
Other Adverse Events (participants affected / at risk) | 14/63 | 4/57
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N-SWEAT Patch (N=63) | Sham Patch (N=57)
Device or Treatment Related Events (Injury, poisoning and procedural complications) | 14 (17) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-04-26): https://cdn.clinicaltrials.gov/large-docs/07/NCT04599907/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-09): https://cdn.clinicaltrials.gov/large-docs/07/NCT04599907/SAP_001.pdf